CLINICAL TRIAL: NCT03591094
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effect of PTI-428 in Subjects With Cystic Fibrosis
Brief Title: Study Assessing PTI-428 Safety, Tolerability, Pharmacokinetics and Effect in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-428-06
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PTI-428 dose level 1 (Active Comparator)
  Interventions: Drug: PTI-428
- PTI-428 dose level 2 (Active Comparator)
  Interventions: Drug: PTI-428
- Placebo PTI-428 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTI-428 — Active
  Arms: PTI-428 dose level 1; PTI-428 dose level 2
Drug: Placebo — Placebo
  Arms: Placebo PTI-428

SUMMARY:
The study population is comprised of adult subjects with cystic fibrosis (CF) who are homozygous for the F508del mutation and are currently receiving background treatment with tezacaftor/ivacaftor for a minimum of 1 month prior to Day 1. The planned sample size is approximately 40 subjects. 20 subjects will be assigned to PTI-428 dose level 1 or placebo and 20 subjects will be assigned to PTI-428 dose level 2 or placebo. At each dose level, subjects will be randomized at a 3:1 randomization ratio. Subjects will receive once daily oral doses of PTI-428 or placebo for 28 days, while the subjects continue to receive background treatment with tezacaftor/ivacaftor per product label. The study drug administration period will be followed by a 14-day safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF with the F508del/F508del genotype on record
* On tezacaftor/ivacaftor dosing for both label indication and per label dosing for a minimum of 1 month on Day 1
* Forced expiratory volume in 1 second (FEV1) 40-90% predicted, inclusive
* Clinically stable with no significant changes in health status within 14 days of Day 1
* Non-smoker and non-tobacco user for a minimum of 28 days prior to screening and for the duration of the study

Exclusion Criteria:

* Participation in another clinical trial or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Study Day 1
* History of cancer within the past 5 years (excluding cervical cancer in situ with curative therapy for at least one year prior to screening and non-melanoma skin cancer)
* History of organ transplantation
* Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness (as determined by the investigator) requiring an increase or addition of medication, such as antibiotics or corticosteroids, within 14 days of Day 1
* Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme®, Cayston®, TOBI®)) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days prior to Day 1
* History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | Baseline through Day 42
  Safety and tolerability will be assessed by adverse events (AEs), safety labs, electrocardiograms (ECGs), physical examinations and vital signs.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
Time of Cmax (Tmax) | 28 days
Area under the concentration time curve from time 0 to time of last measurable concentration (AUC0-t) | 28 days
Change in FEV1 over time | Baseline through Day 42
Change in sweat chloride over time | Baseline through Day 42

OTHER OUTCOMES:
Change in nasal epithelial CFTR mRNA and protein expression over time | Baseline through Day 42
Change in CFQ-R over time | Baseline through Day 42
Cmax of PTI-428 metabolites, if applicable | 28 days
Tmax of PTI-428 metabolites, if applicable | 28 days
AUC0-t of PTI-428 metabolites, if applicable | 28 days

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Stanford University, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - Northwestern University, Chicago, Illinois
  - Cystic Fibrosis Center, Children's Hospital of Illinois at OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Iowa, Roy J and Lucille A Carver College of Medicine, Iowa City, Iowa
  - Universitey of Louisville, Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan Medicine, University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Manchester, New Hampshire
  - Mount Sinai Beth Israel, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Science Center at Tyler - Center for Clinical Research, Tyler, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No